CLINICAL TRIAL: NCT02802449
Title: An Eight Week Double Blinded Randomized, Placebo-controlled Trial to Assess the Effect of Two Doses of 100,000 IU Vitamin D3 by Mouth on Select Genetic Responses in Overweight, Hypertensive African-Americans With Hypovitaminosis D
Brief Title: To Study the Nutri-Genomic Response of Vit-D Supplementation in African-Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: Morehouse School of Medicine (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, David Martins, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-08-2333; 7U54MD008149 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-06-16 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Hypovitaminosis D
Keywords: Vitamin D; Hypovitaminosis D; HTN
MeSH Terms: conditions — Vitamin D Deficiency | interventions — hydroxide ion; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The participant will be randomized to receive two tablets of Placebo (microcrystalline cellulose) to take under direct observation at the baseline and week 2 visit.
  Interventions: Drug: Placebo
- 25 hydroxy-Vitamin D3 or [25 (OH) D3] (Active Comparator): The participant will be randomized to receive two 50,000 IU tablets of oral Vitamin D3 [also known as cholecalciferol or 25 hydroxy-Vitamin D3 or 25 (OH) D3] to take under direct observation at the baseline and week 2 visit.
  Interventions: Drug: 25 Hydroxy- Vitamin D3 [25 (OH) D3]

INTERVENTIONS:
Drug: 25 Hydroxy- Vitamin D3 [25 (OH) D3] — Two 50,000 IU tablets of oral Vitamin D3 [also known as cholecalciferol or 25 hydroxy-Vitamin D3 or 25 (OH) D3] will be given at baseline and 2 weeks after the baseline visit under direct observation by the nurse or research coordinator.
  Other Names: Vitamin D3
  Arms: 25 hydroxy-Vitamin D3 or [25 (OH) D3]
Drug: Placebo
  Arms: Placebo

SUMMARY:
Three hundred thirty (330) overweight, pre-hypertensive/controlled hypertensive, African-American participants will be enrolled in a 8 week study to assess the effect of two administrations of Vitamin D3 on Vitamin D serum responsiveness as a function of clinical, biologic and genetic factors. The investigators anticipate that at least 300 participants will complete this study.

Written, signed and dated informed consent to participate in the study will be given by the participant or a legally acceptable representative, in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related activities/procedures. The original signed and dated consent will be kept in the subject's research file and a copy given to the subject. A copy will also be placed in their medical record.

DETAILED DESCRIPTION:
DETAILED DESCRIPTION OF STUDY PROCEDURES. Three hundred thirty (330) overweight, pre-hypertensive/controlled hypertensive, African-American participants will be enrolled in a 8 week study to assess the effect of two administrations of Vitamin D3 on Vitamin D serum responsiveness as a function of clinical, biologic and genetic factors. The investigators anticipate that at least 300 participants will complete this study.

Written, signed and dated informed consent to participate in the study will be given by the participant or a legally acceptable representative, in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related activities/procedures. The original signed and dated consent will be kept in the subject's research file and a copy given to the subject. A copy will also be placed in their medical record.

BLOOD PRESSURE CONTROL. Controlled high blood pressure is entry criteria, but not an outcome. However, the investigators want to exclude potential participants who are likely to have poor BP control during the study. Therefore, although patients with pre-hypertension or hypertension are eligible to be entered into the study, the protocol only allows enrollment of participants with well-controlled hypertension as defined by SBP≥ 120 mmHg or DBP ≥ 80 mmHg if not on treatment, and SBP <160 mmHg or DBP < 100 mmHg regardless of whether on treatment or not. BP care will be managed by the participants' primary or other provider. All participants being actively treated for hypertension with pharmacotherapy will receive direction to adhere to their medication and to follow-up with their Primary Care Physician. Patients with poorly controlled diabetes as defined by hemoglobin A1c > 8.5% or advanced kidney disease as defined by eGFR < 45 ml/min are excluded. After the study is concluded, all participants will be encouraged and supported to address issues of diet and exercise that may reduce their risk for hypertension. If BP medications need to be adjusted, participants will be referred back to their Primary Care Physician.

VISIT 1 - SCREENING. The screening period will allow for the determination of appropriateness of each subject's inclusion in the study. Written informed consent from the subject or their legally authorized representative would have been obtained prior to any study-related procedures being performed. In addition to signing the general informed consent, subjects who agree to participate the sub-study with fat biopsy will sign a second informed consent.

The subject will be assigned a screening number and will be contacted regarding eligibility once all screening procedures have been performed and laboratory results received.

The following evaluations and assessments will be performed during Screening:

inclusion/exclusion criteria, medical history (including demographics and concomitant medications, including prescription, herbal/vitamins, and all over-the-counter medications), vital signs (sitting BP, heart rate), and a mini physical examination (which will include height (cm), weight (kg), and waist circumference (cm) from which body mass index (BMI) will be calculated and a clinical heart/lung examination. Blood will be drawn (15 cc) for full biochemistry panel with glucose (mg/dl), complete blood count, HbA1c (%), calcium (mg/dl), phosphorus (mg/dl), albumin (mg/dl), pregnancy test and 25(OH)D (ng/ml) levels. After screening information is reviewed and deemed to be appropriate for inclusion in the study, eligible subjects will be given an appointment and preparatory instructions for Visit 2 (Baseline/Randomization/Dose#1). Instructions include cessation of smoking (if they smoke), eating, or drinking caffeine for at least 8 hours prior to the Baseline Visit. If participants are taking prescribed medications, they will be asked to bring them and advised to take them as prescribed.

VISIT 2 - BASELINE/ RANDOMIZATION/ STUDY DRUG DOSE#1 ADMINISTRATION. If subject meets all of the inclusion/exclusion criteria, they will be randomized. The participant will be asked about any adverse events and changes in medications, including prescription, herbal/vitamin, and over-the-counter medications. Vital signs (sitting BP, heart rate) will be obtained and a nutritional survey administered. Blood will be drawn (45 cc) for serum calcium (mg/dl), phosphorus (mg/dl), albumin (mg/dl), iPTH (pg/ml) and 1-84 PTH/7-84 PTH ratio, pregnancy test, 25(OH)D (ng/ml) levels; and samples stored for bio-markers (e.g. pro-inflammatory/pro-thrombotic/fibrotic, insulin sensitivity, and vitamin D receptor polymorphisms). Spot urine sample (30cc) will be collected for calcium/creatinine and albumin/creatinine ratios as well as sodium and isoprostanes. The fat biopsy will be performed on those that agree to be part of the subgroup. Participants undergoing the fat biopsy will be given post biopsy instructions including a return appointment in 7-10 days.

Visit will last about 30-60 minutes for most participants. At the end of the visit, participant will be randomized and given either two 50,000 IU tablets of oral Vitamin D3 [also known as cholecalciferol or 25 hydroxy-Vitamin D3 or 25 (OH) D3] or two tablets of Placebo (microcrystalline cellulose) to take under direct observation. All the participants will be given an appointment and preparatory instructions for Study Visit 3. They will also be asked to avoid any other vitamin D supplements during study period.

VISIT 3 - STUDY DRUG DOSE#2 ADMINISTRATION (2 weeks after baseline). Visit will last about 15 minutes for most participants. Participant will be asked about any adverse events and changes in medications, including prescription, herbal, and over-the-counter medications. Vital signs will be obtained. Participant will be given their second dose of either two 50,000 IU tablets of oral Vitamin D3 or two tablets of Placebo to take under direct observation. All the participants will be given an appointment and preparatory instructions for Study Visit 4 (Week 6).

VISIT 4 (Week 6). During this visit participant will be asked about any adverse events including possible symptoms of vitamin D overdose and changes in medications, including prescription, herbal, and over-the-counter medications. In addition, the following evaluations and assessments will also be performed: vital signs (sitting BP, heart rate). Blood will be drawn (3 tablespoon or 45 cc) for full biochemistry panel, with glucose (mg/dl), HbA1c (%), complete blood count, calcium (mg/dl), phosphorus (mg/dl), albumin (mg/dl), iPTH (pg/ml) and 1-84 PTH/7-84 PTH ratio, and 25(OH)D (ng/ml) levels; and stored samples for bio markers (e.g. pro-inflammatory/pro- thrombotic/fibrotic, insulin sensitivity, and vitamin D receptor polymorphisms). Spot urine sample will be collected for calcium/creatinine and albumin/creatinine ratios as well as sodium and isoprostanes. Urine pregnancy test will also be done. Participants undergoing the fat biopsy will be given post biopsy instructions and will have an additional 7-10 days of follow-up.

VISIT 5 - END OF STUDY (Week 8). At the End of Study visit (EOS), participant will be asked about any adverse events including possible symptoms of vitamin D overdose. In addition, the following evaluations and assessments will also be performed: vital signs (sitting BP and heart rate). The results of the labs from the previous visit will be discussed and if there are any abnormal lab values, participant will be referred to primary care physician for further management.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18-70 years of age and self-identified as African-American or Black
* Pre-hypertension or hypertension (well controlled - see below)
* If a potential study patient is not on treatment their SBP must be > 120 mmHg, or DBP > 80 mmHg
* Whether on treatment or not SBP must be <160 mmHg and DBP must be < 100 mmHg (BP is not an outcome. Controlled BP is for participant safety)
* Screening Vitamin D (D2 and D3 level) >5 and < 25 ng/ml (recommended normal level is > 30 ng/ml)
* Body mass index (BMI) > 25 kg/m2 and < 45 kg/m2
* Any female of non-childbearing potential, including any female who:

  * has had a hysterectomy,
  * has had a bilateral oophorectomy,
  * has had a bilateral tubal ligation or
  * is postmenopausal (demonstration of total cessation of menses for ≥ 1 year prior to the date of the screening visit)
* Any female of child-bearing potential must agree to use at least one form of contraception (may be a barrier method), during the full duration of the study.

Exclusion Criteria:

* Concurrent Disease:

  * Poorly controlled high blood pressure (SBP ≥160 mmHg or DBP ≥ 100 mmHg)
  * Poorly controlled diabetes (HbA1c >8.5%)
  * Screening Vitamin D (D2 and D3 level) < 5 or > 25 ng/ml (recommended normal level is > 30 ng/ml)
  * Estimated glomerular filtration rate (eGFR) < 45 ml/min
  * Evidence of disease that could result in hypercalcemia
  * History of kidney stones (less than one year prior to screening)
  * History of drug, alcohol, or illicit substance abuse (within the past 6 months)
  * History of another chronic disease which the investigator feels should preclude the subject from entering the study (e.g. cancer, immunologic disorder)
  * Liver function tests (LFTs) greater than twice the upper limit of normal
  * Subjects requiring chronic use of nonsteroidal anti-inflammatory drugs or aspirin >325 mg/day
  * Subjects requiring treatment with other vitamin D preparations containing more than 400 IU of vitamin D
  * Subjects requiring chronic use of immunosuppressive therapy or corticosteroids
  * Recent (<6 months) myocardial infarction, stroke, or hospitalization for congestive heart failure
  * Subjects with clinically apparent hypothyroidism or thyrotoxicosis
  * Allergy/intolerance: known allergy to oral vitamin D or microcrystalline cellulose
  * Any female of child-bearing potential who declines to use some method of birth control during the study period

Other:

* Concurrent participation in other clinical trials or taking experimental medications or within 30 days of completing another trial or study.
* Patients who are unable to give informed consent
* Patients who, in the opinion of the Investigator, have a condition which would interfere with their evaluation (e.g. severe mental health disorder)
* Patients who, in the opinion of the Investigator, may experience an unacceptable health risk by participating in this study
* Patients who are pregnant or lactating
* Not African- American or Black by self-identification
* Body mass index (BMI) > 45 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Martins, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The participant will be randomized then given two tablets of Placebo (microcrystalline cellulose) to take under direct observation at the baseline and week 2 visit.
  Placebo
- 25 Hydroxy-Vitamin D3 or [25 (OH) D3]: The participant will be randomized then given two 50,000 IU tablets of oral Vitamin D3 [also known as cholecalciferol or 25 hydroxy-Vitamin D3 or 25 (OH) D3] to take under direct observation at the baseline and week 2 visit.
  25 Hydroxy- Vitamin D3 [25 (OH) D3]: Two 50,000 IU tablets of oral Vitamin D3 [also known as cholecalciferol or 25 hydroxy-Vitamin D3 or 25 (OH) D3] will be given at baseline and 2 weeks after the baseline visit under direct observation by the nurse or research coordinator.
Period: Overall Study
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Started | 111 | 219
Completed | 102 | 202
Not Completed | 9 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3] | Total
Number analyzed (Participants) | 111 | 219 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (9.7) | 51.3 (9.7) | 52.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 91 | 194 | 285
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 111 | 219 | 330
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 219 | 330

OUTCOME MEASURES:

1. Primary Outcome: Plasma PTH Level
Description: Building upon our hypothesis above, this aim exploits the fact that the nuclear Vit-D Receptor (VDR) regulates parathyroid hormone (PTH) gene transcription. Therefore the plasma PTH level serves as a sensitive biomarker of the Vit-D nutri-genomic response. This aim will define the multivariate determinants (covariates such as age, BMI, baseline Vit-D level and dietary calcium) of the Vit-D-PTH level relationship (the primary outcome variable) in African-Americans. It is anticipated that the Vit-D supplementation trial will document a wide variance of Vit-D-PTH level relationships that will identify patients at the upper and lower quartiles of the distribution that are either 'nutrient-responsive' or 'nutrient-resistant'. These studies should help identify the 'clinical' characteristics of the sub-set of African-Americans that exhibit the poorest response to Vit-D supplementation.
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
pg/ml
  Baseline | 58.29 (23.82) | 60.73 (26.04)
  Week 6 | 57.88 (22.23) | 54.05 (26.12)

2. Primary Outcome: Vitamin D3 Level
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
ng/ml
  Baseline | 17.02 (4.51) | 16.55 (4.87)
  Week 6 | 16.64 (4.90) | 32.73 (7.14)

3. Secondary Outcome: Oxidative Stress Markers: Cysteine
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
umol/L
  Cysteine (Baseline) | 253.5 (41.5) | 252.4 (35.6)
  Cysteine (Week 6) | 249.0 (38.7) | 241.2 (32.8)

4. Secondary Outcome: Oxidative Stress Markers: Homocysteine
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
umol/L
  Homocysteine (Baseline) | 11.5 (3.3) | 11.9 (6.1)
  Homocysteine (Week 6) | 11.0 (3.0) | 11.8 (4.8)

5. Secondary Outcome: Oxidative Stress Markers: GSH
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
umol/L
  GSH (Baseline) | 4.1 (1.2) | 4.1 (1.1)
  GSH (Week 6) | 3.6 (0.9) | 3.5 (0.8)

6. Secondary Outcome: Oxidative Stress Markers: Isoprostane
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
Number analyzed (Participants) | 111 | 219
pg/ml
  Isoprostane (Baseline) | 8298.6 (8504.8) | 11914.9 (17904.9)
  Isoprostane (Week 6) | 687.1 (54460.2) | 9979.7 (8630.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout duration of study = 12 weeks.
Arm/Group | Placebo | 25 Hydroxy-Vitamin D3 or [25 (OH) D3]
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/219
Serious Adverse Events (participants affected / at risk) | 1/111 | 0/219
Other Adverse Events (participants affected / at risk) | 5/111 | 15/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | 25 Hydroxy-Vitamin D3 or [25 (OH) D3] (N=219)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | 25 Hydroxy-Vitamin D3 or [25 (OH) D3] (N=219)
Elevated Blood Pressure (Cardiac disorders) | 1 (2) | 4 (5)
Abnormal Lab Value (Renal and urinary disorders) | 0 (0) | 1 (1)
Fractured Right Arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neck Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin Injury - Right Lower Extremity (Pre-Existing) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (2)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back Pain Exacerbation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (2)
Left Shoulder Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash on Bilateral Lower Extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No